CLINICAL TRIAL: NCT06399380
Title: Immediate Effect of Manual Mobilization of the Carpal Bones on the Neural Conduction of the Median Nerve in Patients With Carpal Tunnel Syndrome: Randomized Clinical Trial
Brief Title: In Patients With Carpal Tunnel Syndrome, Median Nerve Conduction is Evaluated After Moving the Wrist Bones
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Elena Bueno Gracia, Physiotherapist, PhD, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI23-440
Record Dates: First submitted 2024-04-25; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual mobilization group (Experimental): Manual mobilization of the carpal bones
  Interventions: Other: Manual mobilization of the carpal bones.
- Placebo group (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Manual mobilization of the carpal bones. — The mobilization of the carpal bones will be done in the following way: patient in supine position, with elbow flexion of approximately 90º, so that the forearm and wrist are almost vertical. The examiner positions the thumb on the dorsal aspect of the scaphoid and trapezius, and the index finger on the dorsal aspect of the piriformis and hamate. Next, a manual ventral force is applied until the resistance of the wrist tissues is felt for 30 seconds. The technique will be repeated 5 times, with a 10-second rest between each application.
  Arms: Manual mobilization group
Other: Placebo — A technique will be performed that will have no effect; the hands will be placed at a point that will not be the carpal tunnel, such as the forearm.
  Arms: Placebo group

SUMMARY:
The goal of this clinical trial is to analyze the immediate effect of manual mobilization techniques of the carpal bones on the median nerve, in patients with carpal tunnel syndrome. The main question it aims to answer is whether there is an immediate positive effect on the electrophysiological variables of the median nerve in patients with carpal tunnel syndrome after performing this technique.

Participants will undergo a carpal bone mobilization technique. There will be a comparison group that will not undergo the technique. The researchers will compare the control and intervention groups to see if the technique has an immediate positive effect.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years
* Present carpal tunnel syndrome diagnosed by electroneurogram
* Have understanding and communication skills
* Give consent to participate in the study.

Exclusion Criteria:

* Having received previous surgery on the hand or wrist
* Present limitation of movement of the carpal bones.
* Not signing the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-05-10 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Distal motor latency (APB) (ms) | Before and immediately after the intervention
Motor amplitude (APB) (mV) | Before and immediately after the intervention
Median motor velocity (m/s) | Before and immediately after the intervention
Median sensory (digit II) (13 cm) (m/sec) | Before and immediately after the intervention
Sensory amplitude (μV ) | Before and immediately after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolny T, Saulicz E, Linek P, Shacklock M, Mysliwiec A. Efficacy of Manual Therapy Including Neurodynamic Techniques for the Treatment of Carpal Tunnel Syndrome: A Randomized Controlled Trial. J Manipulative Physiol Ther. 2017 May;40(4):263-272. doi: 10.1016/j.jmpt.2017.02.004. Epub 2017 Apr 8. PMID 28395984
- [Background] Kim DH, Marquardt TL, Gabra JN, Shen ZL, Evans PJ, Seitz WH, Li ZM. Pressure-morphology relationship of a released carpal tunnel. J Orthop Res. 2013 Apr;31(4):616-20. doi: 10.1002/jor.22271. Epub 2012 Nov 26. PMID 23184493
- [Background] Marquardt TL, Gabra JN, Li ZM. Morphological and positional changes of the carpal arch and median nerve during wrist compression. Clin Biomech (Bristol). 2015 Mar;30(3):248-53. doi: 10.1016/j.clinbiomech.2015.01.007. Epub 2015 Jan 31. PMID 25661267
- [Background] Atroshi I, Gummesson C, Johnsson R, Ornstein E, Ranstam J, Rosen I. Prevalence of carpal tunnel syndrome in a general population. JAMA. 1999 Jul 14;282(2):153-8. doi: 10.1001/jama.282.2.153. PMID 10411196
- [Background] Bueno-Gracia E, Ruiz-de-Escudero-Zapico A, Malo-Urries M, Shacklock M, Estebanez-de-Miguel E, Fanlo-Mazas P, Caudevilla-Polo S, Jimenez-Del-Barrio S. Dimensional changes of the carpal tunnel and the median nerve during manual mobilization of the carpal bones. Musculoskelet Sci Pract. 2018 Aug;36:12-16. doi: 10.1016/j.msksp.2018.04.002. Epub 2018 Apr 4. PMID 29635191
- [Background] Padua L, Coraci D, Erra C, Pazzaglia C, Paolasso I, Loreti C, Caliandro P, Hobson-Webb LD. Carpal tunnel syndrome: clinical features, diagnosis, and management. Lancet Neurol. 2016 Nov;15(12):1273-1284. doi: 10.1016/S1474-4422(16)30231-9. Epub 2016 Oct 11. PMID 27751557
- [Background] Jimenez Del Barrio S, Bueno Gracia E, Hidalgo Garcia C, Estebanez de Miguel E, Tricas Moreno JM, Rodriguez Marco S, Ceballos Laita L. Conservative treatment in patients with mild to moderate carpal tunnel syndrome: A systematic review. Neurologia (Engl Ed). 2018 Nov-Dec;33(9):590-601. doi: 10.1016/j.nrl.2016.05.018. Epub 2016 Jul 22. English, Spanish. PMID 27461181
- [Background] Ibrahim I, Khan WS, Goddard N, Smitham P. Carpal tunnel syndrome: a review of the recent literature. Open Orthop J. 2012;6:69-76. doi: 10.2174/1874325001206010069. Epub 2012 Feb 23. PMID 22470412
- [Background] Newington L, Harris EC, Walker-Bone K. Carpal tunnel syndrome and work. Best Pract Res Clin Rheumatol. 2015 Jun;29(3):440-53. doi: 10.1016/j.berh.2015.04.026. Epub 2015 May 27. PMID 26612240
- [Background] Bueno-Gracia E, Perez-Bellmunt A, Lopez-de-Celis C, Shacklock M, Salas-Lopez A, Simon M, Alvarez-Diaz P, Tricas-Moreno JM. Dimensional changes of the carpal tunnel and median nerve during manual mobilization of the carpal bones - Anatomical study. Clin Biomech (Bristol). 2018 Nov;59:56-61. doi: 10.1016/j.clinbiomech.2018.09.001. Epub 2018 Sep 3. PMID 30195102
- [Background] Jimenez-Del-Barrio S, Cadellans-Arroniz A, Ceballos-Laita L, Estebanez-de-Miguel E, Lopez-de-Celis C, Bueno-Gracia E, Perez-Bellmunt A. The effectiveness of manual therapy on pain, physical function, and nerve conduction studies in carpal tunnel syndrome patients: a systematic review and meta-analysis. Int Orthop. 2022 Feb;46(2):301-312. doi: 10.1007/s00264-021-05272-2. Epub 2021 Dec 3. PMID 34862562

DOCUMENTS (1):
  • Informed Consent Form (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/80/NCT06399380/ICF_000.pdf